CLINICAL TRIAL: NCT01376154
Title: Special Drug Use Investigation for ZEFIX (Lamivudine) Tablet (HBV Cirrhosis)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112335
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed lamivudine tablet: Subjects with hepatitis B virus-induced liver cirrhosis prescribed lamivudine tablet during study period
  Interventions: Drug: Lamivudine

INTERVENTIONS:
Drug: Lamivudine

SUMMARY:
The purpose of this study is to confirm efficacy and safety when administering lamivudine tablet alone in subjects with hepatitis B virus-induced liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with hepatitis B virus-induced liver cirrhosis, in whom lamivudine tablet was administered alone for 6 months or longer, or those in whom lamivudine tablet was expected to be administered alone for 6 months or longer

Exclusion Criteria:

* Subjects previously enrolled in Drug Use Investigation or Special Drug Use Investigation of lamivudine tablet
* Subjects with a history of hypersensitivity of the ingredients of lamivudine tablet

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with hepatitis B virus-induced liver cirrhosis, in whom lamivudine tablet was administered alone for 6 months or longer, or those in whom lamivudine tablet was expected to be administered alone for 6 months or longer.
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse events in Japanese subjects with hepatitis B virus-induced liver cirrhosis treated with lamivudine tablet | 6 months or more

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline